CLINICAL TRIAL: NCT05476965
Title: A Phase II Trial of Cisplatinum, Paclitaxel, and Sintilimab Induction Therapy Followed by De-escalation Radiotherapy for Patients With Postoperative Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Selected De-escalation Radiotherapy for Postoperative Head and Neck Squamous Cell Carcinoma
Acronym: iCSDeR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yu Qian, Doctor, Hubei Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN010815
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Radiotherapy; Immunotherapy; Surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): De-escalation radiation following induction therapy and surgery Drug: Cisplatinum Drug: Paclitaxel Drug: Sintilimab Surgery: Surgery Radiation: De-escalation radiotherapy
  Interventions: Combination Product: induction therapy; surgery; radiotherapy
- Arm 2 (Active Comparator): Arm 2 Standard radiation following induction therapy and surgery Drug: Cisplatinum Drug: Paclitaxel Drug: Sintilimab Surgery: Surgery Radiation: Standard radiotherapy
  Interventions: Combination Product: induction therapy; surgery; radiotherapy

INTERVENTIONS:
Combination Product: induction therapy; surgery; radiotherapy — Radiotherapy: de-escalation radiotherapy or standard radiotherapy

SUMMARY:
This study is looking to see if sintilimab, an anti-PD-1 McAb given with cisplatinum and paclitaxel (2 chemotherapy agents) during induction therapy in advanced head and neck squamous cell carcinoma can significantly shrink the subject's cancer, then de-escalation radiotherapy can be used.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 to 65.
2. Newly diagnosed pathologically confirmed locally advanced head and neck squamous cell carcinoma, including oral cancer, oropharyngeal cancer, laryngeal cancer, while nasopharyngeal carcinoma was excluded. The P16 status of oropharyngeal carcinoma is known.
3. Locally advanced resectable head and neck tumors (stage III and stage IV) were enrolled and radiotherapy is expected to be performed within 4 or 6 weeks after surgery. Tumor staging is based on AJCC/UICC 8th Edition. All the patients must undergo the following examinations to determine the tomor stage before the treatment: complete medical history, physical examination, blood and biochemical routine, head and neck CT or MRI, chest CT scan, abdominal ultrasound and bone scan. In addition, 18F PET/CT can be used to replace the last three imaging examinations mentioned above.
4. ECOG performance status 0 or 1.
5. Normal Organ function

   1. Leukocytes ≥ 4×109/L
   2. Hemoglobin ≥ 90 g/L
   3. Platelets ≥ 100×109/L
   4. Total bilirubin ≤ 1.5x upper limit of normal
   5. Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) ≤ 2.5x upper limit of normal
   6. Alkaline phosphatase ≤ 2.5x upper limit of normal
   7. Creatinine clearance > 60 mL/min
6. Normal thyroid function, amylase, pituitary function, inflammation and infection index, myocardial enzyme, and ECG. For patients with abnormal ECG or cardiovascular history but not meet the exclusion criteria, a cardiac color ultrasound is needed, and the results should be normal.
7. Patients must sign an informed consent form prior to study entry and they must be willing to comply with the visit, treatment protocol, laboratory examination and other requirements included in the study protocol.
8. Women of childbearing potential and men with fertility partners must agree to follow instructions for methods of contraception (such as condoms or contraceptive drugs) from screening to 1 years after completing treatment.

Exclusion Criteria:

1. Positive HBsAg and HBV DNA > 1×103 copies/ml, or anti-HCV antibody positive.
2. Positive anti-HIV antibody or diagnosed as AIDS.
3. patients with active tuberculosis history (whether treated or not) in the past 1 years, or with a history of tuberculosis more than 1 years (except those who had received regular anti-tuberculosis treatment).
4. Has active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary diseases, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Type I diabetes, hypothyroidism requiring hormone replacement therapy, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia) are not included.
5. Diagnosis of interstitial pneumonia or pneumonia and receiving oral or intravenous steroid therapy in the past 1 year.
6. Receiving systemic glucocorticoid (10 mg prednisone per day) therapy or any other form of immunosuppressive therapy (excluding inhaled or topical corticosteroids).
7. Uncontrolled heart disease, such as: heart failure, NYHA level ≥ 2; instability Angina pectoris; myocardial infarction history in the past 1 year; supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
8. Pregnant or breastfeeding female patients (women of childbearing potential must have urine pregnancy test).
9. Suffering from other malignant tumors at previously or currently. Additionally, well treated non melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer are not included.
10. Allergic to macromolecular protein or any component of anti-PD1 antibody.
11. Active infection requiring systemic therapy no more than one week.
12. Has received a live vaccine within 30 days before administrating anti-PD-1 antibody.
13. organ transplantation history.
14. Other situations assessed by the investigator that may endanger patient safety or compliance, such as serious diseases requiring treatment (including mental diseases), serious abnormal test results, or with other family or social high-risk factor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 3 weeks
  pCR was defined as the absence of histologically identifiable residual cancer in any resected specimen. The objective is to intensify induction chemotherapy with the addition of anti-PD-1 McAb sintilimab aimed at acquiring a higher postoperative pCR.

SECONDARY OUTCOMES:
Radiation dose of normal organs and treatment-related adverse events | 12 months
  Assess the radiation dose of normal organs between the de-escalation radiotherapy group or standard radiotherapy group. Furthermore, toxicities reaction between two groups also been compared. Adverse events were any untoward medical occurrence in a participant who received study interventions without regard to possibility of causal relationship.
Safety of sintilimab in combination with chemotherapy | 12 months
  Evaluate the safety of sintilimab in combination with chemotherapy followed by surgery and radiotherapy in advanced head and neck squamous cell carcinoma patients.
Functional assessment of cancer therapy scale head and neck quality of life assessments | 6 months after the use of anti-PD-1 McAb sintilimab
  Evaluate quality of life in all patients. The specific modules H&N35 in Quality of Life Questionnaire Core 30 module (QLQ-C30) and European Organization for Research and Treatment of Cancer (EORTC) and Functional Assessment of Cancer Therapy (FACT) H&N V4.0 were used. Both of them are standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score.
Progression free survival (PFS) in 2 years | 24 months
  PFS was defined as the time from the date of randomization to the first documentation of objective progressive disease (PD) per modified RECIST v1.1 as assessed by Investigator or death (due to any cause), whichever occurred first. Comparing the PFS at 24 months after completing chemotherapy, surgery, and radiotherapy between arm 1 and arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Desheng Hu, Dr., Study Chair — Hubei Cancer Hospital
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China